CLINICAL TRIAL: NCT03782012
Title: Knowledge Accessibility and Availability in Forming Knowledge to Text Inferences Among Middle Grade Readers
Brief Title: Knowledge Accessibility and Availability in Forming Knowledge-to-Text Inferences Among Middle Grade Readers
Acronym: BVU-R15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buena Vista University (Other)
Responsible Party: Principal Investigator, AMY BARTH, Assistant Professor, Buena Vista University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: R15HD092922 (NIH)
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Reading Problem
Keywords: Reading Comprehension; Adolescents; Knowledge Availability and Accessibility; Inference Making
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This study will randomly select 300 from Storm Lake students in grades 5-8 (i.e., 75 students per grade) (see Table 1). Because of the short duration of the experiment (3 sessions), we estimate 20% attrition (n = 60 students). We will replace all students who exit from the sample within grade to ensure sufficiently power. Students will randomly be assigned within grade to one of two conditions: support versus no support.
Who Masked: Participant, Outcomes Assessor
Masking Description: Provide information about other parties who may be masked in the clinical trial,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knowledge Supported (Experimental): Students will have 30 seconds to view pictures of the knowledge base items and discuss relations among items.
  Interventions: Behavioral: Supported
- Knowledge Not Supported (Experimental): Students will be provided 30 seconds to view pictures of the knowledge base items.
  Interventions: Behavioral: Supported

INTERVENTIONS:
Behavioral: Supported — Visual organization of knowledge base items plus discourse-based discussion supporting knowledge availability and accessibility

SUMMARY:
Recent adolescent-based research shows that inference making improves across grades 6-12, uniquely accounts for variance in sentence- and passage-level comprehension, and that individual differences in inference making relate in a principled way to variations in reading comprehension for readers of all abilities (Barth et al., 2015; Barnes et al., 2015). These findings suggest that comprehension requires inference making and that comprehension fails when readers do not possess relevant knowledge (i.e., availability) or slowly retrieve (i.e., accessibility) and integrate knowledge from text or semantic memory during reading (Kendeou, 2015). To date, only one study has examined the effects of knowledge availability and accessibility on inference making among adolescents. To extend this limited body of research, this project will conduct two experimental studies designed to examine (a) the extent to which knowledge-base availability and accessibility relates to the accuracy and rate of constructing inferences using that knowledge (Aim 1) and (b) the extent to which retrieval practice (i.e., spaced practice testing) increases knowledge availability and accessibility and improves the accuracy and rate of forming inferences using that knowledge-base among middle grade readers (Aim 2). In addition, this project will integrate investigative research into an undergraduate Honors Research Program by developing an investigative laboratory component that engages undergraduates in conducting applied research (Aim 3). The research design uses 558 students in grades 5-8. To address Aim 1, mixed effects explanatory item response models will fit to the trial-by-trial reading accuracy and speed data. Repeated measures analysis of variance models will address Aim 2 with analysis of variance models used for Aim 3. The expected outcomes of the proposed research include (a) understanding how knowledge availability and accessibility relate to inference making among adolescent readers; (b) understanding the sources of inference making difficulty; and (c) methods for improving knowledge availability and accessibility and inference making to broadly implement in secondary grade classrooms.

DETAILED DESCRIPTION:
This project conducts experimental studies with three objectives: (1) To determine the extent to which variations in knowledge availability and accessibility influence the rate and accuracy of forming inferences. (2) To investigate whether individual difference factors are potential sources of variability in explaining inference making and reading comprehension. (3)To determine whether systematic retrieval practice improves both knowledge availability and accessibility as well as the accuracy and rate of forming inferences using the knowledge-base. Study 1 Overview. Procedures modify those used by Barnes et al. (1996). In Phase 1, students learn a knowledge-base of 14 facts about Gan. In Phase 2, students will read and listen to an informational text that consists of six sections. A computer asks students comprehension questions that tap information from that text section and the taught knowledge base. Phase 3 retests retention of the knowledge-base. One week later, Phase 4 retests the knowledge-base and students take a larger test battery. All students will complete Phases 1-4 individually. Study participants (n = 300) will come from Storm Lake Community School District students in grades 5-8 (n = 657) with both males and females recruited for participation. The school district will provide demographic data, reading scores from the Iowa Assessment for Reading, and Gates MacGinities Reading Test for all participants from which the investigator will randomly select students for the treatment or control group. The investigator will replace students who exit the sample with students from the same grade who consented but not randomly selected for participation. Participation will exclude students with significant cognitive impairments who participate in the Life Skills Class (e.g., severe autism, behavior, cognitive disability) due to task demands. Additional Assessments measure the constructs of reading comprehension, inference making, word reading efficiency, metacognition, working memory, and background knowledge. Multiple measures of each construct allow the study to identify (a) relations among latent abilities; (b) role of these latent abilities in establishing reading comprehension, independent of measure-specific factors or measurement error; and (c) individual differences that lead to variation in performance. Data Analysis. The investigator will screen for missing data and outliers and evaluate the distributional properties of observed variables, making transformations as necessary and appropriate. If possible, the investigator will correlate non-plausible values or list them as missing if not possible, and label extreme data points. Power. General recommendations on sample sizes in structural equation modeling (SEM) suggest minimum samples of 300 (i.e., 75 participants per grades 5-8). This sample size will allow the research team to detect correlations among constructs greater than 0.05 and regression coefficients in latent variable regressions of 0.05 with over 80% power. Consideration of Biological Variables. To sufficiently power the study and generalize findings, this study recruits males and females for participation and collects gender, race, disability status, and socioeconomic status to determine if these child-attributes moderate knowledge accessibility and availability. Analytic Approach. The investigator will model the effects of knowledge availability and accessibility on inference making without dichotomizing the distribution of comprehension. To determine whether reader characteristics (i.e., knowledge availability and accessibility, metacognition, reading comprehension, word reading efficiency, background knowledge, working memory, and grade) make unique contributions to inference making, the investigator will fit mixed effects explanatory item response models to the trial-by-trial inference making accuracy and speed data with item-level accuracy and reading speeds cross-classified between persons and items. The investigator will also nest people within grade, treating grouping variables for people such as grade and items (i.e., literal, word-to-text, and knowledge-to-text inferences) as fixed factors. If limited variability exists in accuracy data, the investigator will only model response time data. The investigator will also evaluate how organization of knowledge relates to knowledge accessibility and inference making. Structural equation modeling will evaluate relations among the constructs (i.e., comprehension, word efficiency, inference making, knowledge accessibility and availability, metacognition, and working memory) to determine the role of knowledge accessibility and availability in reading comprehension and factors influencing knowledge accessibility and availability. Using Cain et al. (2001) framework, the investigator will classify each inference failure as (1) incorrect text-premise recall (i.e., the participant fails to retrieve the relevant premise from the text); (2) incorrect knowledge-based recall (i.e., the participant fails to retrieve the relevant premise from the knowledge-base); and (3) integration failure (i.e., the participant fails to integrate text content with knowledge). A traditional two-way ANOVA (skill group X inference type) on the incorrect inference response will occur with skilled readers defined as achieving proficiency on the Iowa Assessment for Reading and performance above a standard score of 90 on the Gates MacGinitie Reading Test. The investigator will only compare the means for skilled versus less skilled readers. The investigators hypothesize that: (1) less skilled middle grade readers will make more errors than skilled readers; (2) less skilled readers will not always recognize the need to form inferences during reading relative to skilled readers; and (3) no significant differences will exist across the middle grades (Ahmed et al., 2016; Barth et al., 2015; Barnes et al., 2015). Results of Aim 1 will tell us if less skilled readers need the duration of retrieval practice increased to achieve similar benefits as more skilled readers and if less skilled readers need help organizing the taught knowledge-base so that it is more available and accessible when reading informational texts, which will inform Aim 2 - To examine the extent to which retrieval practice (i.e., spaced practice testing) increases knowledge availability and accessibility and improves the accuracy and rate of forming inferences using that knowledge-base among middle grade readers. Study 2 uses procedures modified from those used by Butler (2010). In Phase 1, students learn a knowledge-base of 14 facts about Gan. In Phase 2, students read and study the six-section informational texts with reassessment of the student's retention of the knowledge base immediately after studying these 6 texts. In Phase 3, students restudy two of the text sections (restudy passages), repeatedly take the same test on another two text sections (same test), and repeatedly take different tests on the other two text sections (variable test). Immediately after interacting with all six text sections, the project reassesses the retention of the knowledge base. Phase 4 occurs one week later and again reassesses the students' retention of the knowledge-base and administers the same additional test battery as in Aim 1. Study participants (n = 180) will come from Storm Lake Community School District students in grade 5-8. The investigators anticipate that students will come from diverse socio-economic and ethnic backgrounds. Student Selection and Exclusions. In the fall of 2019, laboratory assistants will recruit students and screen them with the Gates-MacGinitie Reading Test. Students selected for participation: (1) perform below a standard score of 90 on the Gates-MacGinitie Reading Test; (2) did not participate in Aim 1; and (3) are not enrolled in life skills classes (i.e., severe Autism, behavior, cognitive impairments) due to task appropriateness. The investigator will document any additional services that students receive (i.e., Title, special education, and reading support) and included them as contextual variables in later analyses. Power and Design. The investigators estimate the sample associated with an effect size of 0.25, alpha 0.05, and with over 80% power at 136 participants for between group differences, 36 for within group differences, and 180 for the interaction. Randomization will occur within grade, with all qualified students in grade 5 available for randomization because these students did not participate in Aim 1. The investigators estimate attrition to be 20% or 36 participants total and will replace participants who exit the pool of consented students not randomly selected for participation. Consideration of Biological Variables. To sufficiently power the study and generalize findings, the study recruits males and females for participation and collects gender, race, disability status, and socioeconomic status to determine if these child-attributes moderate knowledge accessibility and availability. Data Analysis. As in Aim 1, the investigators will screen for missing data and outliers and evaluate the distributional properties of observed variables, making transformations as necessary and appropriate. When possible, investigators will correct non-plausible values or listed them as missing if investigators cannot correct them and label extreme data points. Analytic Approach. Data analysis will use repeated measures analysis of variance models to examine the effect of the experimental condition on knowledge retention. Separate ANOVAs will analyze scores obtained on the question types (i.e., explicit text-, word-to-text- and inference-questions) and the different error types by condition. Results of Aim 2 (and Aim 1) and additional analyses will inform the independent research projects conducted by undergraduate laboratory assistants (Aim 3). Aim 3. To integrate investigative research into an undergraduate Honors Research Program. This proposal will support the development of a laboratory component for the Honors Proposal Seminar. This sophomore-level seminar focuses on the organizational structure of their research proposal (i.e., introduction, hypotheses, and method section). The laboratory component will provide students hands-on experiences in the practices of conducting applied research in the schools. Students will also have access to extant data to examine interesting questions related to the reading and reading-related skills of adolescents which should heighten student interest and enthusiasm for conducting research among adolescents. Laboratory Outline. This project will create a two-semester laboratory course (e.g., 32 sessions) that meets weekly for two hours. Lab sessions will address Institutional Review Board applications; appropriate engagement with school personnel; subject recruitment; parent/guardian consent; child assent; formation of research questions and hypotheses; fidelity of implementation; experimental design; inputting and verifying data; analyzing data; and discussing, reporting, and publishing findings (i.e., manuscripts, presentations, and spoken posters). Throughout the year, students will also engage in the primary literature, culminating with the eventual submission of a primary journal article that includes appropriate introduction, method, results, and discussion.

ELIGIBILITY:
Inclusion Criteria:

- Must be able to hear study directions and stimuli

Exclusion Criteria:

* Students who are enrolled in a Life Skills class focused on activities of daily living
* Students who are enrolled in English as a Second language introductory classes
* Students with severe disabilities that impact reading and listening.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 241 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AMY E BARTH, PHD, Principal Investigator — Buena Vista University
Locations (1):
- Storm Lake Community School District, Storm Lake, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All data and related materials are available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: All data and related materials are available upon request.
Access Criteria: All data and related materials are available upon request.

REFERENCES:
- [Background] Barnes MA, Dennis M, Haefele-Kalvaitis J. The effects of knowledge availability and knowledge accessibility on coherence and elaborative inferencing in children from six to fifteen years of age. J Exp Child Psychol. 1996 Apr;61(3):216-41. doi: 10.1006/jecp.1996.0015. PMID 8636665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in the K12 schools.
Pre-assignment Details: Recruitment was significantly influenced by COVID 19 school closures and restrictions that prevented the recruitment of students spring 2020 through the end of the project.
Groups:
- English Language Learners: Participants who reported a home language other than English
- Monolingual English Speakers: Participants who reported English as their primary home language.
Period: Overall Study
Arm/Group | English Language Learners | Monolingual English Speakers
Started | 145 | 96
Cohort 1 | 87 | 58
Cohort 2 | 58 | 38
Completed | 145 | 96
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- English Learners: Students identified, by the school district, as learning English as a second language.
- Monolingual English Speaking Students: Students identified, by the school district, as speaking English as their primary language.
- Total: Total of all reporting groups
Arm/Group | English Learners | Monolingual English Speaking Students | Total
Number analyzed (Participants) | 145 | 96 | 241
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 145 | 96 | 241
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 43 | 122
  Male | 66 | 53 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 89 | 32 | 121
  Not Hispanic or Latino | 53 | 62 | 115
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 37 | 9 | 46
  Native Hawaiian or Other Pacific Islander | 9 | 4 | 13
  Black or African American | 7 | 8 | 15
  White | 0 | 41 | 41
  More than one race | 89 | 32 | 121
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 145 | 96 | 241
FastBridge Adaptive Reading [Mean (Standard Deviation); unit: units on a scale] — FastBridge Adaptive Reading (aReading) is a computer- administered assessment. The aReading test measures students' proficiency in various reading-related domains such as concepts of print, vocabulary, and comprehension of literary and informational text.
  aReading Scaled Score Benchmark: Grade 5: >=523 = College pathway, <509 = some risk, <497 = High risk Grade 6: >=530 = College pathway, <516 = some risk, <502 = High risk
  aReading scores are listed according to bands of 50 points each starting at 350 and ending at max 750. Note this is an extended scale score.
  units on a scale | 510.8 (26.4) | 521.7 (17.5) | 515.14 (23.89)

OUTCOME MEASURES:

1. Primary Outcome: Change in Knowledge Accessibility and Availability
Description: Know-It task is an individually administered assessment of knowledge accessibility (rate of response) and availability (accuracy of response) for a taught knowledge base.
  Scale title is the Know-It, the minimum value is 0 the maximum value is 14, a score of 14 is a better outcome.
  Construct: Literal and Inferential Comprehension Higher score indicates better reading proficiency
Time Frame: immediately after training KNOW-IT knowledge base items; one week after training KNOW-IT knowledge base items; and 1 month after training KNOW-IT knowledge base items
Population: English learners and Monolingual English speaking students (n = 241)
Measure: Mean (Standard Deviation); unit: score on a scale (0 to 14)
Arm/Group | English Learners | Monolingual English Speaking Students
Number analyzed (Participants) | 145 | 96
score on a scale (0 to 14)
  Time 1 immediately after training | 13.2 (1.4) | 13.7 (1.1)
  Time 2 one week after training | 12.28 (2.59) | 13.50 (3.22)
  Time 3 one month after training | 11.65 (2.68) | 12.60 (2.31)

2. Secondary Outcome: Direct and Indirect Effect of Reading Comprehension for Grade Level Texts on Knowledge Accessibility & Availability
Description: Gates-MacGinite Reading Test-4th Edition, a standardized, group-administered, multiple-choice assessment of reading comprehension with internal consistency for students in grades 5-8 that exceeds 0.80. The scale title is the Gates-MacGinitie Test 4th Edition, Reading Comprehension subtest. Higher score means a better outcome.
  Standard score with a mean of 100 and standard deviation of 15. Standard score range from 55 to 145.
  Data on this measure was only collected for Cohort 1 (n = 145) and not for Cohort 2 (n = 96)
  Construct: Reading Comprehension Higher score indicates better reading proficiency
Time Frame: 180 days from training of KNOW-IT knowledge base items
Population: Data on this measure was only collected for Cohort 1 (n = 145) and not for Cohort 2 (n = 96) Population Analyses (Cohort 1 only) = 145 (87 English learners + 58 Monolingual English Speaking students)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | English Learners | Monolingual English Speaking Students
Number analyzed (Participants) | 87 | 58
score on a scale | 103 (9.4) | 106 (9.4)

3. Secondary Outcome: Direct and Indirect Effect of Reading Strategy Use for Content Area Texts on Knowledge Availability and Accessibility
Description: Contextualized Reading Survey, students to report study strategies used when reading. The scale measures the types of reading strategies readers use in different types of reading situations. For each question, the reader indicates their use on a scale of 1 to 5. 1 means I almost never do this. 2 means that I rarely do this. 3 means that I sometimes to this. 4 means that I usually do this. 5 means that I almost always do this. Items load onto 4 factors: evaluation and knowledge integration; pragmatic strategies; self regulation; help seeking. Higher values indicate a better outcome.
  Toal of 49 items on the survey. Min score 49 max score 245.
  Construct: Strategic reading skills
Time Frame: 45 days from training of KNOW-IT knowledge base items
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | English Learners | Monolingual English Speaking Students
Number analyzed (Participants) | 143 | 96
score on a scale | 159.92 (30.70) | 145.72 (25.23)

4. Secondary Outcome: Direct and Indirect Effect of Word and World Knowledge and Understanding on Knowledge Accessibility and Availability
Description: Kauffman Brief Intelligence Test-2, Verbal Knowledge subtest is a norm-referenced, individually administered assessment of expressive word and world knowledge. Internal consistency ranges from 0.89-0.94 for students in grades 5-8.
  Standard score with a mean of 100 and standard deviation of 15. Standard score range from 55 to 145.
  Construct: Vocabulary and verbal knowledge Higher score indicates better vocabulary and verbal knowledgeproficiency
Time Frame: 180 days from training of KNOW-IT knowledge base items
Population: 241
Measure: Mean (Standard Deviation); unit: Units on a Standard Score
Arm/Group | English Learners | Monolingual English Speaking Students
Number analyzed (Participants) | 145 | 96
Units on a Standard Score | 89.9 (14.5) | 96.1 (11.8)

5. Secondary Outcome: Direct and Indirect Effect of Reading Fluency for Words on Knowledge Accessibility and Availability
Description: Test of Word Reading Efficiency-2 Sight Word Efficiency, a 45-second assessment of students' word reading accuracy and speed. Reliability coefficients exceed .80 for students in grade 5-8.
  Standard score with a mean of 100 and standard deviation of 15. Standard score range from 55 to 145.
  Construct: Word reading or Decoding skills Higher score indicates better word reading skills
Time Frame: 180 days from training of KNOW-IT knowledge base items
Population: 241
Measure: Mean (Standard Deviation); unit: Units on a Standard Score
Arm/Group | English Learners | Monolingual English Speaking Students
Number analyzed (Participants) | 145 | 96
Units on a Standard Score | 89.2 (27.4) | 90.46 (23.13)

6. Secondary Outcome: Direct and Indirect Effect of Text to Text Inference Making on Knowledge Accessibility and Availability
Description: Bridge-IT, a computerized task, asks students to read a five-sentence text, form an inference, and determine if the next provided sentence continues the story. Internal consistency for students in the middle grades ranges from 0.83-0.87.
  Students were asked to respond to 20 inferential questions. Min score 0, max score 20.
  Higher score indicates better outcome. Construct: Inference making
Time Frame: 45 days from training of KNOW-IT knowledge base items
Population: Due to severe missingness this data has not been analysed yet.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | English Language Learners | Monolingual English Speakers
Number analyzed (Participants) | 108 | 66
units on a scale | 12.1 (4.02) | 13.9 (4.35)

7. Secondary Outcome: Direct and Indirect Effect of Nonverbal Reasoning on Knowledge Accessibility and Availability
Description: Kauffman Brief Intelligence Test-2 Matrices subtest assess students nonverbal reasoning and ability to identify patterns and problem solve. Reliability coefficients exceed .80 for students in grades 5-8.
  Standard score with a mean of 100 and standard deviation of 15. Standard score range from 55 to 145.
  Construct: Nonverbal reasoning skills Higher score indicates better Nonverbal reasoning skills
Time Frame: 45 days from training of KNOW-IT knowledge base items
Population: 241
Measure: Mean (Standard Deviation); unit: Units on a Standard Score
Arm/Group | English Learners | Monolingual English Speaking Students
Number analyzed (Participants) | 145 | 96
Units on a Standard Score | 98.2 (15.3) | 106.5 (12.1)

8. Secondary Outcome: Direct and Indirect Effect of Working Memory for Words on Knowledge Accessibility and Availability
Description: Working Memory Test from the Woodcock Johnson. This subtest measures students' memory for numbers.
  Standard score with a mean of 100 and standard deviation of 15. Standard score range from 55 to 145.
  Construct: Working memory Higher score indicates better working memory capacity
Time Frame: 45 days from training of KNOW-IT knowledge base items
Population: 234
Measure: Mean (Standard Deviation); unit: Units on a Standard Score
Arm/Group | English Learners | Monolingual English Speaking Students
Number analyzed (Participants) | 143 | 91
Units on a Standard Score | 98.0 (14.8) | 100.8 (17.0)

9. Secondary Outcome: Test of Word Reading Efficiency Sight Word Reading. Construct: Word Reading
Description: Assesses students speed of reading words by sight.
  Scores reported are standard scores with a mean of 100 and standard deviation of 15 Standard score range from 55 to 145.
  Construct: Word reading or decoding skills Higher score indicates better word reading skills
Time Frame: 45 days from training of KNOW-IT knowledge base items
Population: 234
Measure: Mean (Standard Deviation); unit: Units on a Standard Score
Arm/Group | English Language Learners | Monolingual English Speakers
Number analyzed (Participants) | 143 | 91
Units on a Standard Score | 97.06 (12.58) | 100.91 (11.20)

10. Secondary Outcome: Direct and Indirect Effect of Working Memory for Text on Knowledge Accessibility and Availability
Description: Woodcock Johnson Verbal Memory task requires that the student listen to a series of words and determine if the words have been heard before.
  Standard score with a mean of 100 and standard deviation of 15. Standard score range from 55 to 145.
  Construct: Verbal working memory Higher score indicates better verbal working memory capacity
Time Frame: 45 days
Population: 234
Measure: Mean (Standard Deviation); unit: Units on a Standard Score
Arm/Group | English Learners | Monolingual English Speaking Students
Number analyzed (Participants) | 143 | 91
Units on a Standard Score | 95.8 (18.9) | 99.6 (19.3)

11. Secondary Outcome: Direct and Indirect Effect of Reading Fluency for Nonwords on Knowledge Accessibility and Availability
Description: Test of Word Reading Efficiency-2, Phonemic Decoding Efficiency, a 45-second assessment of students' non-word reading accuracy and speed. Alternate form reliability exceeds 0.90 for students in grades 5-8.
  Standard score with a mean of 100 and standard deviation of 15 Standard score range from 55 to 145.
  Construct: Decoding or word reading skills Higher score indicates better word reading skills
Time Frame: 45 days from training of KNOW-IT knowledge base items
Population: 234
Measure: Mean (Standard Deviation); unit: Units on a Standard Score
Arm/Group | English Language Learners | Monolingual English Speakers
Number analyzed (Participants) | 143 | 91
Units on a Standard Score | 97.80 (13.70) | 100.22 (12.68)

12. Secondary Outcome: Direct and Indirect Effect of Reading Fluency for Connected Text on Knowledge Accessibility and Availability
Description: Curriculum Based Measure of Oral Reading Fluency, is an assessment of students ability to read connected text quickly and accurately. Reliability coefficients exceed .80 for students in grades 5-8.
  Scores represent the average number of words read correctly on the oral reading fluency assessment.
  Higher score indicates better word reading fluency skills
  Construct: Reading fluency
Time Frame: 180 days from training of KNOW-IT knowledge base items
Measure: Mean (Standard Deviation); unit: words read correctly
Arm/Group | English Learners | Monolingual English Speaking Students
Number analyzed (Participants) | 87 | 58
words read correctly | 167 (22.6) | 168 (23.2)

13. Secondary Outcome: Direct and Indirect Effect of Reading Comprehension for Grade Level Texts on Knowledge Accessibility and Availability
Description: FastBridge Adaptive Reading (aReading) is a computer adaptive assessment of reading comprehension. Reliability coefficients exceed .80 for students in grades 5-8. The aReading test measures students' proficiency in various reading-related domains such as concepts of print, vocabulary, and comprehension of literary and informational text.
  aReading Scaled Score Benchmark: Grade 5: >=523 = College pathway, <509 = some risk, <497 = High risk Grade 6: >=530 = College pathway, <516 = some risk, <502 = High risk
  aReading scores are listed according to bands of 50 points each starting at minimum 350 and ending at maximum 750. Note, this is an extended scale score.
  Construct: Reading skills
Time Frame: 180 days from training of KNOW-IT knowledge base items
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | English Learners | Monolingual English Speaking Students
Number analyzed (Participants) | 145 | 96
score on a scale | 510 (22.3) | 519 (18.6)

14. Secondary Outcome: Direct and Indirect Effect of Word, World, and Domain Knowledge on Knowledge Accessibility and Availability
Description: Gates MacGinitie Reading Test Vocabulary subtest measures students understanding of word, world, and domain knowledge using multiple choice questions. Reliability coefficients exceed .80 for students in grades 5-8
  Standard score with a mean of 100 and standard deviation of 15. Standard score range from 55 to 145.
  Construct vocabulary knowledge Higher score indicates better vocabulary knowledge
Time Frame: 180 from training of KNOW-IT knowledge base items
Population: 145
Measure: Mean (Standard Deviation); unit: Units on a Standard Score
Arm/Group | English Learners | Monolingual English Speaking Students
Number analyzed (Participants) | 87 | 58
Units on a Standard Score | 99 (9.2) | 100 (10.0)

ADVERSE EVENTS:
Time Frame: Up to 1 school year for each participant.
Description: Adverse events were not anticipated with this project. However, adverse events were systematically assessed in two ways. First, parental informed consent and child assent was obtained prior to testing. If a child refused to participate, they did not participate. Second, we regularly met with the school principal to obtain adverse event information from the perspective of the school district.
Arm/Group | English Learners | Monolingual English Speaking Students
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/96
Other Adverse Events (participants affected / at risk) | 0/145 | 0/96

LIMITATIONS AND CAVEATS:
The sample was relatively small, and results of this study are based on a sample of students from one rural school district. Data was collected from one cohort of typically developing readers and one cohort of at-risk readers across two years and combined for our primary and secondary analyses. Next, we were unable to administer or did not have access to students' scores on multiple measures due to restrictions related to COVID-19. Third, students with significant disabilities were excluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT03782012/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT03782012/ICF_001.pdf